CLINICAL TRIAL: NCT04933422
Title: Phase 1 Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Effects of CM93 in Subjects With Recurrent Glioblastoma (rGBM) Characterized by Epidermal Growth Factor Receptor (EGFR) Mutation or Amplification
Brief Title: CM93 Treatment in Subjects With Epidermal Growth Factor Receptor (EGFR)-Modified Recurrent Glioblastoma (rGBM)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Crimson Biopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CM93-101
Record Dates: First submitted 2021-05-24; First posted 2021-06-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Glioblastoma
Keywords: EGFR; rGBM; EGFR-altered rGBM
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CM93 pre-treatment arm (Experimental): Applicable only for part 3 of this trial (surgical window of opportunity), pre-treatment with CM93 prior to surgical resection of recurrent glioblastoma
  Interventions: Drug: CM93
- No pre-treatment arm (No Intervention): Applicable only for part 3 of this trial (surgical window of opportunity), no pre-treatment prior to surgical resection of recurrent glioblastoma

INTERVENTIONS:
Drug: CM93 — oral capsule of CM93 administered once daily
  Other Names: N-(5-((4-(1H-pyrrolo[2,3-b]pyridin-1-yl)pyrimidin-2-yl)amino)-2-((2-(dimethylamino)ethyl)(methyl)amino)-4-methoxyphenyl)acrylamide 4-methylbenzenesulfonate
  Arms: CM93 pre-treatment arm

SUMMARY:
This is a first-in-human study of CM93, an oral investigational drug, in adults with Epidermal Growth Factor Receptor-modified glioblastoma. The study is designed in three parts consisting of a dose-escalation phase, a dose-expansion phase and a window-of-opportunity surgical trial. The trial objectives are to evaluate the safety, pharmacokinetics, pharmacodynamics and clinical effects of CM93 in this patient population.

DETAILED DESCRIPTION:
CM93 is a third-generation, covalent/irreversible, brain penetrant small molecule Epidermal Growth Factor Receptor (EGFR) tyrosine kinase inhibitor. It is not a substrate of p-glycoprotein or breast cancer resistance protein (bcrp) and is a mild inhibitor of bcrp. It is a potent inhibitor of EGFR mutations but also has activity against wild type EGFR.

This first-in-human phase I trial will evaluate the safety, tolerability, and pharmacokinetics (PK) of CM93 and determine the recommended Phase 2 dose (RP2D) for further evaluation using a 3+3 design (Part 1). Once the RP2D has been determined 12 additional patients will be treated in a dose expansion cohort to confirm the safety and tolerability of the selected dose (Part 2). Subsequent to the phase I trial a window-of-opportunity surgical trial will initiate. Tumor from both contrast enhancing and non-contrast enhancing areas of patients who received CM93 before surgery will be resected and evaluated to determine if therapeutic concentrations of the drug are achieved. Pharmacodynamic studies will be conducted in tumor tissue from patients who received CM93 before surgery and the patients who did not receive drug before surgery to determine if there is adequate inhibition of EGFR. After recovery from surgery all 30 patients will receive CM93 until progression, development of unacceptable toxicity, or withdrawal of consent and preliminary evidence of activity will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed recurrent or progressive World Health Organization IV isocitrate dehydrogenase (IDH) wild type glioblastoma and variants, including high-grade astrocytoma with molecular features of glioblastoma (WHO grade IV).
2. Archival tumor from initial or other prior surgery is documented to have EGFR mutation or EGFR amplification
3. Previous first line therapy with at least radiotherapy utilizing standard dosing of CNS radiation with or without chemotherapy.
4. Patients must have shown unequivocal evidence of tumor progression by MRI and have confirmed measurable disease per RANO criteria.
5. Patients must have confirmation of availability of sufficient tissue from prior surgery revealing glioblastoma or variants for submission following registration for repeat EGFR mutation testing and additional sequencing. The following amount of tissue is required:

   * 1 formalin-fixed paraffin-embedded (FFPE) tumor tissue block (preferred), or
   * 20 FFPE unstained slides (5 µm thickness)
6. Patients must have recovered to grade 0 or 1 as determined by the National Cancer Institute CTCAE version 5.0 or pre-treatment baseline from clinically significant toxic effects of prior therapy (including but not limited to exceptions for alopecia, laboratory values listed per inclusion criterion 3.1.12, and lymphopenia which is common after therapy with temozolomide).
7. An interval of at least 4 weeks (to registration) between prior surgical resection or one week from stereotactic biopsy.
8. Age ≥18 years. Because no dosing or adverse event data are currently available on the use of CM93 in participants <18 years of age, children are excluded from this study, but will may be eligible for future pediatric trials.
9. Karnofsky performance status ≥ 60 (Appendix A).
10. Participants must have adequate organ and marrow function as defined below:

    * absolute neutrophil count ≥1,500/mcL
    * hemoglobin ≥ 9g/dL
    * platelets ≥100,000/mcL
    * total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (subjects with Gilbert syndrome are allowed if direct bilirubin within normal limits)
    * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
    * creatinine ≤1.5mg/dL or a calculated creatinine clearance ≥60mL/min
    * negative serum beta-hCG test in women of childbearing potential (defined as women ≤50 years of age, or >50 years of age with a history of amenorrhea ≤12 months prior to study entry).
11. Left ventricular ejection fraction (LVEF) at least 50% by echocardiogram or multigated acquisition scan (MUGA).
12. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
13. The effects of CM93 on the developing human fetus are unknown. For that reason, women of childbearing age must agree to use dual contraceptive methods which, in the opinion of the principal investigator, are effective and adequate for that subject's circumstances while on study drug and for 4 months afterward.
14. Men who partner with a woman of childbearing potential must agree to use effective, dual contraceptive methods (i.e., a condom, with female partner using oral, injectable or barrier method) while on study drug and for 4 months afterward.
15. Ability to understand and the willingness to sign a written informed consent document.

    Additional criteria for window-of-opportunity surgical cohort
16. Patients must be undergoing surgery for recurrent or progressive disease that is clinically indicated as determined by their care providers.
17. Ability of a neurosurgeon to gross or subtotally resect both enhancing and non-enhancing components of the tumor and that sufficient tissue can be obtained from each component for correlative studies.

Exclusion Criteria:

* 1. Prior evidence of IDH mutation by IHC or DNA sequencing (i.e., IDH wild type only)

  2. Participants who have had prior treatment with any EGFR inhibitor, or VEGF or VEGFR inhibitor.

  3. Participants who have had temozolomide less than 23 days from study initiation, treatment with CCNU or BCNU less than 42 days from study initiation, or treatment with any cancer-directed systemic therapy less than 4 weeks or 5 half-lives from study initiation, whichever is shorter.

  4. Participants who have had any cancer-directed immunomodulatory or molecularly-targeted agent or monoclonal antibody within 14 days prior to initiation of study drug.

  5. Participants who have used any investigational agents within 28 days or 5 half-lives from study initiation, whichever is shorter.

  6. For phase 1 dose escalation and dose expansion: increasing corticosteroid requirement or a dose >6 mg per day of dexamethasone or equivalent dose of other corticosteroids within 7 days prior to study initiation. This does not apply to patients in the window-of-opportunity surgical trial.

  7. Participants who received radiation therapy within 12 weeks prior to registration, unless there is surgical confirmation of recurrent disease or evidence of new enhancing recurrent disease outside of the prior radiotherapy treatment field.

  8. Participants with major surgery within the last 28 days prior to registration.

  9. History of allergic reactions attributed to compounds of similar chemical or biologic composition to CM93.

  10. Participants receiving any medications or substances that are strong inhibitors of CYP3A4 (e.g., clarithromycin, azole antifungals, protease inhibitors, nefazadone, grapefruit juice) or those metabolized by CYP 3A4/3A5 are ineligible. Caution is advised for participants taking dexamethasone as well as strong inducer(s) of its metabolism. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.

  11. Participants with known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness.

  12. Participants with any of the following within 6 months prior to initiation of study drug: uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack.

  13. Pulmonary embolism within 1 month prior to initiation of study drug.

  14. Unstable cardiac dysrhythmias or persistent prolongation of the QTc (Fridericia) interval to >450msec for males or >470msec for females.

  15. Any contraindication to contrast-enhanced MRI examination.

  16. Evidence of Grade ≥ 2 intracranial hemorrhage.

  17. Participants with any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the Investigator's opinion, would make the subject inappropriate for entry into this study.

  18. Participants with uncontrolled intercurrent illness, including active or clinically unstable bacterial, viral or fungal infection requiring systemic therapy.

  19. Pregnant women are excluded from this study; there are no reproductive toxicity data at the stage of development in animals. CM93 may have potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CM93, breastfeeding should be discontinued if the mother is treated with CM93.

  20. Previous malignancy, except for non-squamous cell cancer of the skin or carcinoma in situ of the uterine or cervix, unless the natural history or treatment of the tumor does not interfere with the safety or efficacy assessment of the investigational regimen.

  21. Participants with difficulty swallowing/unable to swallow pills; malabsorption syndrome; refractory nausea and vomiting, chronic gastrointestinal (GI) disease or previous significant bowel resection with clinically significant sequelae that would preclude adequate absorption of study drug.

Additional criteria for window-of-opportunity surgical cohort

22. Participants with >2 prior relapses of glioblastoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | 28 days
  Record and compare safety and tolerability, adverse events, changes in laboratory parameters and electrocardiogram measure of patients to baseline measurements. DLTs (dose-limiting toxicities) are defined as a clinically significant adverse event (AE) or laboratory abnormality unrelated to disease progression that meet certain criteria.
Maximum tolerated dose | 28 days
  The MTD (maximum tolerated dose) is defined as the highest dose level at which ≤1 of 6 subjects experience a DLT during Cycle 1 (the first 28 days of intervention).
Recommended phase 2 dose | 28 days
  Determined by the DSMC (Data Safety Monitoring Committee) after review of safety data, the RP2D (recommended phase 2 dose) will be the MTD unless:
  * Significant clinical anti-tumor effect (complete response, partial response, or stable disease for ≥2 months) is seen below the MTD, in which case a clinically active dose level may be selected as an RP2D; or
  * Toxicities observed beyond Cycle 1 require reducing the RP2D(s) below the MTD level; or
  * MTD is not achieved, in which case the highest dose level administered may become an RP2D.
Concentration of CM93 in non-enhancing areas of tumor | 7 days
  In part 3 of the study, tissue samples from non-enhancing areas of the tumor will be analyzed for CM93 and concentration will be reported for the CM93-treated group.

SECONDARY OUTCOMES:
Half-life of CM93 | 22 days
  Calculate half-life from the plasma bioanalysis of CM93 and its active metabolite at different time points and doses.
Maximum plasma concentration (Cmax) | 22 days
  Calculate Cmax from the plasma bio analysis of CM93 and its active metabolite.
Time to Maximum plasma concentration (Tmax) | 22 days
  Calculate Tmax from the plasma bio analysis of CM93 and its active metabolite.
Area under the curve (AUC) | 22 days
  Calculate AUC from the plasma bio analysis of CM93 and its active metabolite.
EGFR level in tumor specimens | 7 days
  In part 3 of the study, average pEGFR (phosphorylated epidermal growth factor receptor) levels in the tumor specimens of CM93-treated surgical patients will be compared to the levels in tumor specimens from untreated patients and difference between the two groups noted.

IPD SHARING:
Plan to Share IPD: Undecided